CLINICAL TRIAL: NCT07395479
Title: A Phase I Study of the In Vivo CAR-T Platform for Treating Advanced Malignant Tumors Based on Target Screening
Brief Title: A Platform Study of In Vivo CAR-T for Treating Advanced Malignant Tumors Based on Target Screening
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC5276
Record Dates: First submitted 2026-01-10; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Advanced Malignant Tumours
Keywords: in vivo CAR-T; DLL3; GPRC5D; BCMA

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- V001-BCMA (Experimental): Intravenous administration of V001-BCMA as a single agent for patients with B-cell-related hematologic malignancies. Dose cohorts: 1x10^8 TU、2x10^8 TU、≤4x10^8 TU and ≤8x10^8 TU.
  Interventions: Genetic: V001-BCMA
- V001-GPRC5D (Experimental): Intravenous administration of V001-GPRC5D as a single agent for patients with B-cell-related hematologic malignancies. Dose cohorts: 1x10^8 TU、2x10^8 TU、≤4x10^8 TU and ≤8x10^8 TU.
  Interventions: Genetic: V001-GPRC5D
- V001-DLL3 (Experimental): Intravenous administration of V001-BCMA as a single agent for patients with small cell lung cancer. Dose cohorts: 1x10^8 TU、2x10^8 TU、≤4x10^8 TU and ≤8x10^8 TU.
  Interventions: Genetic: V001-DLL3

INTERVENTIONS:
Genetic: V001-BCMA — An in vivo CAR-T drug targeting BCMA administered intravenously
  Arms: V001-BCMA
Genetic: V001-GPRC5D — An in vivo CAR-T drug targeting GPRC5D administered intravenously
  Arms: V001-GPRC5D
Genetic: V001-DLL3 — An in vivo CAR-T drug targeting DLL3 administered intravenously
  Arms: V001-DLL3

SUMMARY:
This is a single-arm, open-label, single-center, dose-escalation Phase I platform study designed to evaluate the safety, tolerability, preliminary efficacy, pharmacokinetics, and pharmacodynamics of an in vivo CAR-T therapy (V001 Injection, targeting BCMA, GPRC5D, DLL3, etc.) in patients with advanced malignant tumors.

DETAILED DESCRIPTION:
This is a single-arm, open-label, single-center, dose-escalation Phase I platform study designed to evaluate the safety, tolerability, preliminary efficacy, pharmacokinetics, and pharmacodynamics of an in vivo CAR-T therapy (V001 Injection, targeting BCMA, GPRC5D, DLL3, etc.) based on a lentiviral vector platform in patients with advanced malignant tumors (including hematological malignancies and solid tumors). The study employs a platform design, enrolling patients into different cohorts based on target and indication.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Histologically confirmed advanced hematological malignancies (e.g., multiple myeloma, lymphoma) or solid tumors (e.g., small cell lung cancer) that are relapsed or refractory.
* Tumor cells express the relevant target (e.g., BCMA, GPRC5D, DLL3) as required for the specific cohort.
* ECOG performance status 0-2 (hematological malignancies) or 0-1 (solid tumors) and life expectancy ≥ 3 months.
* Adequate organ function (e.g., creatinine clearance ≥45 mL/min, LVEF ≥45%).
* Patients of childbearing potential must agree to use effective contraception during the study and for 1 year after dosing.
* Signed informed consent form.

Exclusion Criteria:

* Active, uncontrolled infection.
* Active central nervous system metastases or involvement.
* Prior anticancer therapy, radiotherapy, or investigational therapy within specified timeframes before the first study dose.
* Severe cardiac or pulmonary disease (e.g., NYHA Class III/IV heart failure), severe hepatic or renal impairment.
* Active Hepatitis B, Hepatitis C, HIV, or syphilis infection.
* Prior allogeneic hematopoietic stem cell transplantation (within specified window) or active graft-versus-host disease.
* Pregnancy or lactation.
* History of severe allergy to any components of the investigational product.
* Any other condition deemed by the investigator to increase risk or interfere with study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-11-21 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose-Limiting Toxicities (DLTs) | Within 28 days after the first infusion
  Incidence and characteristics of DLTs graded according to NCI CTCAE v5.0. The DLT observation period is 28 days post-infusion.
Maximum Tolerated Dose (MTD) | During the dose-escalation phase (approximately 12 months)
  To determine the MTD of V001 Injection.
Incidence of Adverse Events (AEs) | From signing ICF until 24 months after the last infusion.
  Incidence and severity of treatment-emergent adverse events (TEAEs) graded according to NCI CTCAE v5.0.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | At Day 28, Months 2, 3, 6, 9, 12, 18, 24 post-infusion
  Best overall response rate assessed per indication-specific criteria.
Duration of Response (DOR) | From date of the first response until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Time from first achieving response to disease progression or death.
Progression-Free Survival (PFS) | From date of infusion until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  From date of infusion until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
Overall Survival (OS) | From the date of infusion until the date of death from any cause, assessed up to 24 months
  Time from infusion to death from any cause
Peak concentration of CAR-T cells in peripheral blood | At multiple timepoints post-infusion up to Month 24
  Peak concentration of CAR-T cells in peripheral blood
time to peak of CAR-T cells in peripheral blood | At multiple timepoints post-infusion up to Month 24
  time to peak of CAR-T cells in peripheral blood
AUC of CAR-T cells in peripheral blood | At multiple timepoints post-infusion up to Month 24
  AUC of CAR-T cells in peripheral blood

OTHER OUTCOMES:
Cytokine levels | At multiple timepoints post-infusion up to Month 24
  Pharmacodynamic Biomarkers
CRP | At multiple timepoints post-infusion up to Month 24
  Pharmacodynamic Biomarkers
Ferritin | At multiple timepoints post-infusion up to Month 24
  Pharmacodynamic Biomarkers
Immunogenicity | Baseline, Day 28, Months 3, 6, 9, 12
  Incidence of anti-drug antibodies.

CONTACTS AND LOCATIONS:
Overall Officials: Shuhang Wang, PhD, Study Director — Clinical Trial Center
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences 17 Panjiayuan Nanli, Chaoyang District, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No